CLINICAL TRIAL: NCT06869434
Title: In Cesarean Sections, is the Length of the Thoracolumbar Vertebral Column Applicable for Determining the Dosage of Bupivacaine in Spinal Anesthesia?
Brief Title: Thoraco Lumbar Vertebral Length and Bupivacaine Dosage in C-Section
Acronym: bupivacaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kudret Dogru, Professor. Dr., TC Erciyes University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/62
Record Dates: First submitted 2025-02-27; First posted 2025-03-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obstetric Anesthesia Problems; Bupivacaine Adverse Reaction
Keywords: Vertebral length, bupivacaine, cesarean,spinal, hypotension
MeSH Terms: conditions — Hypotension | interventions — Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group VBL (Vertebral body length) received 0.2 mg x VBL cm of %0.5 hyperbaric bupivacaine, (Active Comparator): Patients in Group VBL (Vertebral body length) received 0.2 mg x VBL cm of 0.5% hyperbaric bupivacaine
  Interventions: Procedure: Group VBL (Thoracolumbal vertebral body length) received 0.2 mg x VBL cm of %0.5 hyperbaric bupivacaine
- Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated ac (Active Comparator): Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated according to the patient's height 0.065 mg/cm
  Interventions: Procedure: Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated according to the patient's height 0.065 mg/cm
- Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height (Active Comparator): Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight
  Interventions: Procedure: Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight.

INTERVENTIONS:
Procedure: Group VBL (Thoracolumbal vertebral body length) received 0.2 mg x VBL cm of %0.5 hyperbaric bupivacaine — intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight. A dosage was derived using Harten's dose chart formulated for Caucasian parturients
  Other Names: Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated according to the patient's height 0.065 mg/cm
  Arms: Group VBL (Vertebral body length) received 0.2 mg x VBL cm of %0.5 hyperbaric bupivacaine,
Procedure: Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated according to the patient's height 0.065 mg/cm — Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated according to the patient's height 0.065 mg/cm
  Arms: Group FD (fixed dose) received a volume of 0.5% hyperbaric bupivacaine based on a dose calculated ac
Procedure: Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight. — Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight.
  Arms: Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height

SUMMARY:
Our hypothesis is that the bupivacaine dose determined according to the thoracolumbar vertebral body length (VBL) is more effective in achieving a lower hypotension rate during spinal anesthesia for cesarean delivery than the dose usually adjusted based on height and weight. The VBL measurements were determined from the midpoint of C7 to the tuffier line L4 spinous process.

Method: Patients ranging in height from 150 to 170 were randomly assigned to either Group 1 (0.2 mg of 0.5% hyperbaric bupivacaine per cm VBL or Group 2 (height-adjusted dose of 0.5% hyperbaric bupivacaine based on a minimum dose of 0.065 mg/cm according to height) or Group 3 (height-adjusted dose of 0.5% hyperbaric bupivacaine based on a minimum height-adjusted dose of 0.065 mg/cm).

DETAILED DESCRIPTION:
The study followed a parallel study strategy. Patients provided informed permission before the procedure. The study was randomly assigned and blinded. The study was conducted from April 2025 to May 2026. Patients with pre-existing or pregnancy-induced hypertension, cardiovascular or cerebrovascular disease, contraindications to spinal anesthesia, weighing < 50 kg or > 110 kg, and heights higher than 170 cm or shorter than 150 cm were eliminated. Informed written consent was acquired from all patients participating in the trial. Each patient was evaluated for vital parameters and possible complications at 3-minute intervals before and after the spinal anesthesia application, treated if necessary, and recorded. The study was concluded at the end of the cesarean section.

There was no premeditation among the patients. The patient had standard monitoring, including non-invasive blood pressure, ECG, and pulse oximetry, with recorded baseline blood pressure and heart rate measurements. We inserted two 20-gauge intravenous cannulas and administered an IV-balanced solution using these routes. The patients' age, height, weight, ASA class, and VBL (C7-L4 Tuffier line cm) were recorded. The Tuffier's line (TL), which is made by drawing a horizontal line across the tops of the iliac crests, is the most common anatomical landmark right now. It has been shown to match up with the L4-L5 interspace or the L4 spinous process.

After skin infiltration with 2% lidocaine, a 25-gauge short-bevel Quincke spinal needle was placed at the L3-4 vertebral interspace with the patient in a sitting position. After aspiration of cerebrospinal fluid, the following anesthetic solutions were delivered over 5 seconds. Randomization was used to divide the patients into three groups. The trial was double-blind, with the patient and assessor unconscious of their group allocation. Only the practitioner delivering the spinal anesthesia was aware of the group allocation. Systolic, diastolic, and mean arterial blood pressure and heart rate were documented at baseline and assessed at 3-minute intervals, commencing 3 minutes post-spinal injection and persisting until the initiation of surgical procedures, after which measurements were conducted at 3-minute intervals.

Patients in Group VBL (Vertebral Body Length) received 0.2 mg x VBL cm of 0.5% hyperbaric bupivacaine. In contrast, Group FD (fixed dose) received a 0.5% hyperbaric bupivacaine volume based on a dose calculated according to the patient's height of 0.065 mg/cm. Group AD (adjusted dosage) got intrathecal heavy bupivacaine (0.5%) tailored to the patient's height and weight. A dosage was derived using Harten's dose chart formulated for Caucasian parturients

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) Class II
2. Having regular antenatal visits
3. Singleton pregnancy at ≥37 weeks of gestation
4. Pregnant women aged 18-45 -

Exclusion Criteria:

1. Those with eclampsia, those with preeclampsia
2. Undergoing an emergency cesarean section
3. Those with bleeding diathesis and those receiving anticoagulant therapy
4. With a history of carotid artery stenosis,
5. Cardiovascular disease,
6. Hypertension,
7. Chronic obstructive pulmonary disease,
8. Heart rhythm outside of sinus
9. Patients with a history of cerebrovascular disease
10. Alcoholism or psychiatric illness
11. Placenta previa, accreta, and percreta

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 285 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Hypotension rate among the groups | From the patient's arrival in the operating room to the end of the surgery
  Our hypothesis is that the bupivacaine dose determined according to the thoracolumbar vertebral body length (VBL) is more effective in achieving a lower hypotension rate during spinal anesthesia for cesarean delivery than the dose usually adjusted based on height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Kudret Dogru, Prof. Dr., Study Director — TC Erciyes University
Locations (1):
- Kudret Doğru, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui KM, Ali MA, Ullah H. Comparison of spinal anesthesia dosage based on height and weight versus height alone in patients undergoing elective cesarean section. Korean J Anesthesiol. 2016 Apr;69(2):143-8. doi: 10.4097/kjae.2016.69.2.143. Epub 2016 Mar 30. PMID 27066205
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Bower JR, Kinsella SM. Preventing and treating hypotension during spinal anaesthesia for caesarean section. BJA Educ. 2020 Nov;20(11):360-361. doi: 10.1016/j.bjae.2020.08.001. Epub 2020 Sep 9. No abstract available. PMID 33456918
- [Background] Carpenter RL, Caplan RA, Brown DL, Stephenson C, Wu R. Incidence and risk factors for side effects of spinal anesthesia. Anesthesiology. 1992 Jun;76(6):906-16. doi: 10.1097/00000542-199206000-00006. PMID 1599111
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35755061/